CLINICAL TRIAL: NCT04980339
Title: Multimodal Imaging Evaluation and Prognostic Analysis of Participants With Transposition of the Great Arteries After Arterial Switch Operation: a Multi-site Clinical Study
Brief Title: Multimodal Imaging Evaluation and Prognostic Analysis of Participants After Arterial Switch Operation
Status: Not yet recruiting | Type: Observational
Sponsor: Xie Mingxing (Other)
Collaborators: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other); Shanghai Zhongshan Hospital (Other); Henan Provincial People's Hospital (Other); Wuhan Asia Heart Hospital (Other); Guangdong Provincial People's Hospital (Other)
Responsible Party: Sponsor-Investigator, Xie Mingxing, Head of Department of Ultrasound, Union Hospital, Union Hospital, Tongji Medical College, Huazhong University of Science and Technology
Organization: Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other)
Other Study IDs: 2021 ASO V1.0
Record Dates: First submitted 2021-07-10; First posted 2021-07-28 (Actual); Last update posted 2022-07-13 (Actual); Status verified 2022-07

CONDITIONS: Arterial Switch Operation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- ASO group: All participants with TGA/TBA after ASO

SUMMARY:
The aims of this study are to

1. Identify the early and midterm outcomes in terms of mortality and reoperation of the arterial switch operation (ASO).
2. Identifying the influence of coronary artery anomalies on the in-hospital and post-discharge prognosis after ASO.
3. Evaluate the predictors for neoaortic valve regurgitation after ASO.
4. Explore the risk factors for neopulmonary artery stenosis after ASO.

DETAILED DESCRIPTION:
This study will enroll participants with transposition of the great arteries (TGA) and double outlet right ventricle with subpulmonary ventricular septal defect (VSD) (Taussig-Bing anomaly, TBA). The cardiac structure and function will be evaluated by multimodal imaging including transthoracic echocardiographic examination, stress echocardiography, cardiac computed tomography scan, cardiovascular magnetic resonance imaging.

And the study aimed to:

1. Identify the early and midterm outcomes in terms of mortality and reoperation of the arterial switch operation (ASO) in participants with transposition of the great arteries (TGA) and double outlet right ventricle with subpulmonary ventricular septal defect (VSD) (Taussig-Bing anomaly, TBA).
2. Identifying subclinical coronary abnormalities and silent myocardial ischemia by multimodel Imaging, further determine the influence of coronary artery anomalies on the in-hospital and post-discharge prognosis in participants with TGA and TBA after ASO.
3. Evaluate the time course and predictors for neoaortic root dilatation and neoaortic valve regurgitation in participants with TGA and TBA after ASO by multimodel Imaging.
4. Assess the structure of the right ventricular outflow tract and neopulmonary artery in participants with TGA and TBA after ASO by multimodel Imaging, and explore the incidence and risk factors for neopulmonary artery stenosis.

ELIGIBILITY:
Inclusion Criteria:

·Participants with the diagnosis of TGA or TBA underwent ASO.

Exclusion Criteria:

* Patients with various forms of TGA undergoing Réparation à l'Etage Ventriculaire procedure
* Patients with various forms of TGA undergoing Rastelli procedure
* Patients with various forms of TGA undergoing Nikaidoh procedure
* Patients with various forms of TGA undergoing Fontan operation
* Patients with various forms of TGA undergoing atrial repair (Mustard or Senning) operations
* ASO is used as a corrective therapy for prior operations.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All participants diagnosed with TGA or TBA underwent ASO in the hospital with an eligible cardiovascular surgery center.
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2022-10-01 (Estimated); Primary Completion 2032-10-31 (Estimated); Study Completion 2032-10-31 (Estimated)

PRIMARY OUTCOMES:
All cause mortality | Ten years
  Number of participants with all cause mortality after ASO

SECONDARY OUTCOMES:
Cardiac caused mortality | Ten years
  Number of participants with cardiac caused mortality after ASO
All cause reoperation | Ten years
  Number of participants with all cause reoperation after ASO
Right-ventricular outflow tract obstruction and pulmonary branch stenosis | Ten years
  Degree of more than moderate right-ventricular outflow tract obstruction in millimetre of mercury, degree of pulmonary branch stenosis in millimetre of mercury
Neoaortic valve regurgitation | Ten years
  Vena contracta width of neoaortic valve regurgitation in milimetre, ratio of Jet width/LVOT width in percentage

CONTACTS AND LOCATIONS:
Overall Officials: Li Zhang, PhD, Principal Investigator — Department of Ultrasound, Union Hospital, Wuhan, China

IPD SHARING:
Plan to Share IPD: No